CLINICAL TRIAL: NCT05122949
Title: User Satisfaction of Customised 3D Printed Ankle-Foot Orthosis in Comparison to Thermoformed Ankle-Foot Orthosis for Patients With Neurological Conditions: A Preliminary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/00541
Record Dates: First submitted 2021-10-20; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Spinal Cord Injuries; Nerve Palsy
Keywords: 3D print; Digitisation; Ankle-foot orthosis; user satisfaction
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with neurological disorders (Experimental)
  Interventions: Device: 3D Printed Ankle-Foot Orthosis; Device: Thermoformed Ankle-Foot Orthosis

INTERVENTIONS:
Device: 3D Printed Ankle-Foot Orthosis — 3D Printed (Fused Deposition Modelling) Ankle-Foot Orthosis with Polyamide Nylon-12 material
Device: Thermoformed Ankle-Foot Orthosis — Thermoformed Ankle-Foot Orthosis with homopolymer polypropylene

SUMMARY:
Study Design and Subject Recruitment: This was a cross-sectional study in a single centre outpatient setting at the Foot Care and Limb Design Centre, Tan Tock Seng Hospital. As this was a proof-of-concept clinical trial for the introduction of 3D printed AFOs as a patient service, only 5 subjects were recruited based on consecutive sampling.

Interventions: Thermoformed AFOs moulded over the subject's lower limb plaster model served as the control intervention. The plaster models were rectified by an orthotist with over 20 years of experience and the AFO design was determined according to the subject's clinical presentation and needs. The AFOs were manufactured from 4 - 5mm thick homopolymer polypropylene. 3D printed AFOs served as the treatment intervention. It was fabricated through 3D scanning with an Artec Eva 3D scanner (Artec 3D, Luxembourg, Luxembourg) and an adjustable Perspex glass foot plate, CAD modelling with the OrtenShape software (Proteor, Saint-Apollinaire, France), and printed using fused deposition modelling with the Fortus 450mc (Stratasys, Minnesota, United States). The 3D printed AFO is printed of Polyamide Nylon-12 material in the same thickness as the thermoformed AFO. There were no blinding procedures as both interventions were distinctly different and it is not possible to blind subjects with daily use of the AFOs.

Trial Schedule: A thermoformed and a 3D printed AFO were fitted to each subject in a single session. The QUEST survey was administered post-fitting. Subjects brought home both AFOs and were instructed to wear them during ambulation, alternating between the AFOs daily. Subjects returned for follow-up at 3 weeks and 6 weeks post-fitting for necessary adjustments and the administration of the QUEST surveys was repeated for each AFO.

ELIGIBILITY:
Inclusion Criteria:

* Existing patients of the centre,
* Clinical need for an AFO due to neurological disorders.

Exclusion Criteria:

* Cognitive impairment
* Lower limb volume fluctuations
* Severe foot/ ankle varus or valgus deformities
* Lower limb contractures of over 10°
* Non-community ambulators

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) scores | Baseline, 3 weeks follow-up and 6 weeks follow-up
  QUEST 2.0 comprises of 12 items, with 8 items related to user satisfaction with assistive devices and 4 service-related items. Responses for the QUEST items were based on a 5-level response scale, with 1 - Not satisfied at all; 2 - Not very satisfied; 3 - More or less satisfied; 4 - Quite satisfied; and 5 - Very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore